CLINICAL TRIAL: NCT00387218
Title: Exercise, Physical Function, and Parkinson's Disease
Brief Title: Exercise Study For People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD043770 (NIH); COMIRB #02-750
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Parkinson's Disease
Keywords: Exercise; Physical Functional Ability; Spinal Range of Motion; Balance; Economy of Movement; Aerobic Conditioning; Quality of Life; Adherence
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise Therapy

INTERVENTIONS:
Behavioral: Exercise, Physical therapy

SUMMARY:
This study is designed to compare three different exercise approaches to learn which program is best for people with early and mid-stage Parkinson's disease. Results from this study will help determine if participants can maintain the benefits from exercise and will help determine which program people with Parkinson's disease are more likely to continue using.

DETAILED DESCRIPTION:
This is an intervention study that will determine whether an exercise program targeting spinal extremity range of motion for individuals with Parkinson's Disease, is superior to general conditioning and to 'usual care'. This study builds on previous findings of Schenkman and colleagues including the following: loss of spinal and extremity range of motion occur as sequelae to PD; these losses contribute significantly to early impairments of balance; and both spinal range of motion and balance of people with economy of movement is impaired in people who have PD. Specifically, we will examine whether the intervention, targeting range of motion and balance, also improves economy of movement.

Untreated impairments of range of motion, balance, and economy of movement may become highly disabling. Short term improvements of range of motion and balance occur with exercise. If the patient can sustain such improvements after a supervised exercise program is completed, these functionally limiting impairments may be delayed. Additionally, if exercises for spinal range of motion are coupled with functional retraining, the patient should improve in overall physical functional ability. Therefore, this study will establish the overall impact of a targeted exercise program for people with PD in terms of balance, economy of movement, and overall functional ability.

The study is a randomized clinical trial, with three treatment arms and four repeated measures: before treatment, after treatment, and follow-up after 10 months and again after 16 months. This study compares usual care based on the National Parkinson's Foundation, aerobic training, and targeted flexibility and functional training. The primary outcomes are measures of overall functional ability, balance and economy of movement. Secondary outcomes include measures of disease state, spinal range of motion, aerobic capacity, and quality of life.

ELIGIBILITY:
Inclusion Criteria: Community dwelling, independently ambulatory adults with mild to moderate PD (Stages 2, 2.5, and 3 on the modified Hoehn and Yahr scale) will be included. For inclusion, study subjects must have a diagnosis of PD made by their attending neurologist using criteria from the UK Brain Bank (e.g., at least two of the cardinal signs of PD [i.e., bradykinesia, resting tremor, rigidity, postural instability]); without PD medication other known or suspected causes of parkinsonism. They must be on a stable regimen for at least one month prior to enrollment, and must be receiving optimal medication management in the judgment of the examining neurologist.

Exclusion Criteria: Participants will be excluded if: on-state freezing; hospitalized within the previous three months, a score on the Folstein Mini-Mental Status Exam of less than 25 (indicating significant dementia); non-drug induced psychosis, or drug induced hallucinations, off periods of >25% time (UPDRS part IV)[3] or sub-optimal therapy of Parkinson's disease motor or non-motor symptoms; a second neurological disorder (e.g. stroke) with resulting motor involvement, or poorly controlled or unstable cardiovascular disease that precludes participation in the exercise program. In addition, participants will be excluded if they are participating in another trial except for those investigations that meet the following criteria: 1) PD Trial that is not related to the symptoms of PD (e.g., genetics of PD); 2) stable dose of an investigational medication given to treat motor symptoms of Parkinson's disease on an open-label basis or 3) in a trial that is not expected to affect PD or movement (e.g., hypertension, diabetes). They will be excluded if they cannot speak English and do not have adequate interpretation to participate in all aspects of the study.

Other exclusion criteria include presence of atypical parkinsonism syndromes due to drugs (e.g., metoclopramide, flunarizine), metabolic neurogenetic disorders (e.g., Wilson's disease), encephalitis, cerebrovascular, or degenerative disease (e.g. progressive supranuclear palsy, multiple system atrophy, vascular parkinsonism), history of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant. Finally, participants will be excluded if they have any other clinically significant medical condition, psychiatric condition, drug or alcohol abuse, or laboratory abnormality which would, in the judgement of the investigator, interfere with the subject's ability to participate in the study.

Additional exclusions are: 1) exercise limiting neuromuscular, joint/bone, cardiovascular, peripheral vascular, cerebrovascular or pulmonary disease; 2) abnormal treadmill stress test or contraindication to testing (recent MI, CHF, pulmonary embolus, significant aortic stenosis); 3) uncontrolled hypertension; 4) unstable diabetes or other endocrinopathy; 5) active liver disease (>3X normal LFTs); 6) major psychiatric illness that would affect the ability to understand and cooperate fully with the study protocol; 7) massive obesity (BMI>40); anemia; 8) consistent use of alcohol (>2 drinks/d); 9) involvement in an ongoing exercise program (>2Xwk for 20 min at an intensity that could produce sweating) in the last 6 months.

-

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2002-12; Primary Completion 2009-04 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Balance (Functional Reach)
Economy of movement (Oxygen consumption)
Functional capacity (Continuous Scale Physical Functional Performance Test (Cs-PFP)

SECONDARY OUTCOMES:
UPDRS Motor subscale
UPDRS ADL subscale
Quality of life (PDQ-39)
Spinal Range of Motion (Functional Axial Rotation, FAR)
VO2 submax

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Schenkman, PhD, PT, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Waldron's Peak Physical Therapy, Boulder, Colorado
  - Penrose Hospital, Colorado Springs, Colorado
  - University of Colorado at Denver and Health Sciences Center, Denver, Colorado
  - Carmody Recreation Center, Lakewood, Colorado

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886